CLINICAL TRIAL: NCT06121479
Title: Oral Branched-chain Amino Acid Supplementation for Decompensated Cirrhotic Patients: a Pilot Study
Brief Title: Oral Branched-chain Amino Acid Supplementation for Decompensated Cirrhotic Patients
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phunchai Charatcharoenwitthaya, Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI 608/2023
Record Dates: First submitted 2023-11-01; First posted 2023-11-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Decompensated Cirrhosis and Ascites
Keywords: Decompensated cirrhosis; Branched-chain amino acid; Nutrition; Ascites
MeSH Terms: conditions — Ascites | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Intervention Model Description: Oral branched-chain amino acid (BCAA) is provided to the patients with a recommended daily intake of approximately 13.68 grams per day. Each sachet contains 6.84 grams of BCAA (valine 1.82 grams, leucine 3.29 grams, isoleucine 1.72 grams), total protein 17.08 grams, carbohydrates 25.48 grams, fat 5.66 grams, providing 221.2 kcal of energy. Each sachet weighs 52 grams and should be mixed with 150 ml of water. The recommended daily intake is 2 sachets, to be consumed after breakfast and dinner. The BCAA provided to the patients comes in pre-packaged silver sachets, with the manufacturing date and expiration date indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- branched-chain amino acid (Experimental): Oral branched-chain amino acid (BCAA) is provided to the patients with a recommended daily intake of approximately 13.68 grams per day. Each sachet contains 6.84 grams of BCAA (valine 1.82 grams, leucine 3.29 grams, isoleucine 1.72 grams), total protein 17.08 grams, carbohydrates 25.48 grams, fat 5.66 grams, providing 221.2 kcal of energy. Each sachet weighs 52 grams and should be mixed with 150 ml of water. The recommended daily intake is 2 sachets, to be consumed after breakfast and dinner. The BCAA provided to the patients comes in pre-packaged silver sachets, with the manufacturing date and expiration date indicated.
  Interventions: Drug: Branched-chain amino acid

INTERVENTIONS:
Drug: Branched-chain amino acid — Oral branched-chain amino acid is provided to the patients with a recommended daily intake of approximately 13.68 grams per day. Each sachet contains 6.84 grams of BCAA (valine 1.82 grams, leucine 3.29 grams, isoleucine 1.72 grams), total protein 17.08 grams, carbohydrates 25.48 grams, fat 5.66 grams, providing 221.2 kcal of energy. Each sachet weighs 52 grams and should be mixed with 150 ml of water. The recommended daily intake is 2 sachets, to be consumed after breakfast and dinner. The BCAA provided to the patients comes in pre-packaged silver sachets, with the manufacturing date and expiration date indicated.

SUMMARY:
The goal of this clinical trial is to compare the nutritional parameters after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL.

The main questions it aims to answer are:

1. Would thigh muscle thickness change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
2. Would triceps skin fold thickness, mid-arm circumferences, mid-arm muscle circumferences, skeletal muscle mass, appendicular skeletal muscle mass, skeletal muscle index and fat mass change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
3. Would handgrip strength change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
4. Would serum albumin change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
5. Would score for cirrhotic severity such as Model for End-Stage Liver Disease-Sodium Score (MELD-Na score) and Child Turcotte Pugh Score change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?

Participants will be asked to do following tasks:

1. Participants will be asked for basic information such as age, place of residence, and contact telephone number.
2. Participants will undergo measurements of weight, height, body mass index, skinfold thickness on the arms, circumference of the arms and legs, muscle mass, and body fat content using a body composition analyzer, both at the beginning and end of the research study.
3. Participants will perform grip strength measurements, at both the beginning and end of the research study.
4. Participants will undergo laboratory tests, including a complete blood count, liver and kidney function tests, blood clotting factors, and blood mineral levels, with a total blood volume of approximately 15 milliliters (1 tablespoon), collected twice during the study (at the beginning and end).
5. Participants will be administered supplements containing branched-chain amino acids (BCAA) twice a day for a total of 12 weeks.
6. Participants will be appointed for follow-up during the study, totaling 2 appointments at weeks 4 and 12. Side effects related to medication will be asked.
7. Participants will undergo ultrasound measurements of the right thigh to assess thigh muscle thickness, both at the beginning and end of the research study.
8. Participants will will complete questionnaires to assess your overall quality of life twice, both at the beginning and end of the research study.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare the nutritional parameters after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL.

The main questions it aims to answer are:

1. Would thigh muscle thickness change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
2. Would triceps skin fold thickness, mid-arm circumferences, mid-arm muscle circumferences, skeletal muscle mass, appendicular skeletal muscle mass, skeletal muscle index and fat mass change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
3. Would handgrip strength change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
4. Would serum albumin change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?
5. Would score for cirrhotic severity such as Model for End-Stage Liver Disease-Sodium Score (MELD-Na score) and Child Turcotte Pugh Score change after 12-week supplementation of branched-chain amino acids in cirrhotic patients with ascites and serum albumin less than 3 g/dL?

Participants will be asked to do following tasks:

1. Participants will be asked for basic information such as age, place of residence, and contact telephone number.
2. Participants will undergo measurements of weight, height, body mass index, skinfold thickness on the arms, circumference of the arms and legs, muscle mass, and body fat content using a body composition analyzer, both at the beginning and end of the research study.
3. Participants will perform grip strength measurements, at both the beginning and end of the research study.
4. Participants will undergo laboratory tests, including a complete blood count, liver and kidney function tests, blood clotting factors, and blood mineral levels, with a total blood volume of approximately 15 milliliters (1 tablespoon), collected twice during the study (at the beginning and end).
5. Participants will be administered supplements containing branched-chain amino acids (BCAA) twice a day for a total of 12 weeks.
6. Participants will be appointed for follow-up during the study, totaling 2 appointments at weeks 4 and 12. Side effects related to medication will be asked.
7. Participants will undergo ultrasound measurements of the right thigh to assess thigh muscle thickness, both at the beginning and end of the research study.
8. Participants will will complete questionnaires to assess your overall quality of life twice, both at the beginning and end of the research study.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhotic patients of all etiology with aged of 18-85 years
2. Clinically detectable ascites
3. Serum albumin < 3 g/dL

Exclusion Criteria:

1. Patients with hepatocellular carcinoma outside the Milan criteria.
2. Patients with history of gastrointestinal bleeding and spontaneous bacterial peritonitis (SBP) within the last 3 months.
3. Patients with acute on chronic liver failure (ACLF).
4. Patients with uncontrollable chronic comorbidities, including chronic heart failure in NYHA stages 3-4, end stage kidney disease requiring dialysis, and chronic obstructive pulmonary disease Gold D.

5 .Patients who have undergone liver or kidney transplant. 6. Patients with Human Immunodeficiency Virus (HIV). 7. Pregnant or lactating patients. 8. Patients who have undergone large volume paracentesis (>5 liters) with intravenous albumin administration on the day of study enrollment. 9. Patients with a history of above-knee amputation surgery. 10. Patients with a history of receiving intravenous albumin administration every 1-2 weeks within the last one month.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
thigh muscle thickness by ultrasound | 12 weeks
  Thigh muscle thickness (centimeters) by ultrasound of right thigh will be performed according to these instructions 1. Measure the thickness of the right thigh muscles, which are the rectus femoris and vastus intermedius, at a position one-third between the upper edge of the patella bone to the iliac crest, with the patient lying flat. In that position, measure the thigh muscle thickness using two methods: a. Compression reading: Measure the muscle thickness by pressing the probe head until it cannot be compressed further. b. Feather weight reading: Measure the muscle thickness without applying pressure to the probe head. Take the muscle thickness measurements twice for each method, calculate their averages. Increase in thigh muscle thickness implies better nutritional status.
Average Feather Index | 12 weeks
  The Average Feather Index (cm/m2) will be calculated by taking average of thigh muscle thickness (centimeter) measured by feather weight reading divided by height (m^2). Increase in average feather index implies better nutritional status.
Average Compression Index | 12 weeks
  The Average Compression Index (cm/m2) will be calculated by taking average of thigh muscle thickness (centimeter) measured by compression weight reading divided by height (m^2). Increase in average compression index implies better nutritional status.

SECONDARY OUTCOMES:
triceps skin fold thickness | 12 weeks
  Triceps skin fold thickness (TSF, millimeter) will be measured using Lange skin fold caliper at midpoint of non dominant arm.
mid-arm circumferences | 12 weeks
  Mid-arm circumferences (MAC, centimeters) will be measured using standard measuring tape at midpoint of non dominant arm. Increase of mid-arm circumferences implies better nutritional status.
mid-arm muscle circumferences | 12 weeks
  Mid-arm muscle circumferences (MAMC, centimeters) will be obtained from calculating the following formula: MAMC (cm) = MAC - (0.314 × TSF [mm]). Increase of mid-arm muscle circumferences implies better nutritional status.
skeletal muscle mass | 12 weeks
  Skeletal muscle mass (kilograms) will be measured using bioelectrical impedance analysis. Increase of skeletal muscle mass implies better nutritional status.
appendicular skeletal muscle mass | 12 weeks
  Appendicular skeletal muscle mass (kilograms) will be measured using bioelectrical impedance analysis. Increase of appendicular skeletal muscle mass implies better nutritional status.
skeletal muscle index | 12 weeks
  Skeletal muscle index (kilograms/m^2) will be measured using bioelectrical impedance analysis. Increase of skeletal muscle index implies better nutritional status.
Fat mass | 12 weeks
  Fat mass (kilograms) will be measured using bioelectrical impedance analysis.
Handgrip strength | 12 weeks
  Handgrip strength (kilograms) will be measured three times for each hand using digital handgrip strength dynamometer. Increase of handgrip strength implies better physical performance.
MELD Na Score | 12 weeks
  MELD Na Score will be calculated at the start and end of study. Decrease of MELD Na Score implies improving of cirrhotic severity.
Child Turcotte Pugh Score | 12 weeks
  Child Turcotte Pugh Score will be calculated at the start and end of study. Decrease of Child Turcotte Pugh Score implies improving of cirrhotic severity.
Serum albumin | 12 weeks
  Serum albumin (gram/deciliter) will be measured at the start and end of study. Increase of serum albumin implies better nutritional status.

CONTACTS AND LOCATIONS:
Overall Officials: Phunchai Charatcharoenwitthaya, M.D., Principal Investigator — Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand
Locations (1):
- Division of Gastroenterology, Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
In order to protect patients' confidentiality, we will not share individual participant data.

REFERENCES:
- [Background] Liu YB, Chen MK. Epidemiology of liver cirrhosis and associated complications: Current knowledge and future directions. World J Gastroenterol. 2022 Nov 7;28(41):5910-5930. doi: 10.3748/wjg.v28.i41.5910. PMID 36405106
- [Background] D'Amico G, Garcia-Tsao G, Pagliaro L. Natural history and prognostic indicators of survival in cirrhosis: a systematic review of 118 studies. J Hepatol. 2006 Jan;44(1):217-31. doi: 10.1016/j.jhep.2005.10.013. Epub 2005 Nov 9. No abstract available. PMID 16298014
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on nutrition in chronic liver disease. J Hepatol. 2019 Jan;70(1):172-193. doi: 10.1016/j.jhep.2018.06.024. Epub 2018 Aug 23. PMID 30144956
- [Background] Maharshi S, Sharma BC, Srivastava S. Malnutrition in cirrhosis increases morbidity and mortality. J Gastroenterol Hepatol. 2015 Oct;30(10):1507-13. doi: 10.1111/jgh.12999. PMID 25974421
- [Background] Soeters PB, Fischer JE. Insulin, glucagon, aminoacid imbalance, and hepatic encephalopathy. Lancet. 1976 Oct 23;2(7991):880-2. doi: 10.1016/s0140-6736(76)90541-9. PMID 62115
- [Background] Tajiri K, Shimizu Y. Branched-chain amino acids in liver diseases. Transl Gastroenterol Hepatol. 2018 Jul 30;3:47. doi: 10.21037/tgh.2018.07.06. eCollection 2018. PMID 30148232
- [Background] Gluud LL, Dam G, Les I, Marchesini G, Borre M, Aagaard NK, Vilstrup H. Branched-chain amino acids for people with hepatic encephalopathy. Cochrane Database Syst Rev. 2017 May 18;5(5):CD001939. doi: 10.1002/14651858.CD001939.pub4. PMID 28518283
- [Background] Hernandez-Conde M, Llop E, Gomez-Pimpollo L, Fernandez Carrillo C, Rodriguez L, Van Den Brule E, Perello C, Lopez-Gomez M, Abad J, Martinez-Porras JL, Fernandez-Puga N, Ferre C, Trapero M, Fraga E, Calleja JL. Adding Branched-Chain Amino Acids to an Enhanced Standard-of-Care Treatment Improves Muscle Mass of Cirrhotic Patients With Sarcopenia: A Placebo-Controlled Trial. Am J Gastroenterol. 2021 Nov 1;116(11):2241-2249. doi: 10.14309/ajg.0000000000001301. PMID 34074812
- [Background] Siramolpiwat S, Limthanetkul N, Pornthisarn B, Vilaichone RK, Chonprasertsuk S, Bhanthumkomol P, Nunanan P, Issariyakulkarn N. Branched-chain amino acids supplementation improves liver frailty index in frail compensated cirrhotic patients: a randomized controlled trial. BMC Gastroenterol. 2023 May 15;23(1):154. doi: 10.1186/s12876-023-02789-1. PMID 37189033
- [Background] Haj Ali S, Abu Sneineh A, Hasweh R. Nutritional assessment in patients with liver cirrhosis. World J Hepatol. 2022 Sep 27;14(9):1694-1703. doi: 10.4254/wjh.v14.i9.1694. PMID 36185724
- [Background] Sirisunhirun P, Bandidniyamanon W, Jrerattakon Y, Muangsomboon K, Pramyothin P, Nimanong S, Tanwandee T, Charatcharoenwitthaya P, Chainuvati S, Chotiyaputta W. Effect of a 12-week home-based exercise training program on aerobic capacity, muscle mass, liver and spleen stiffness, and quality of life in cirrhotic patients: a randomized controlled clinical trial. BMC Gastroenterol. 2022 Feb 14;22(1):66. doi: 10.1186/s12876-022-02147-7. PMID 35164698
- [Background] Tandon P, Low G, Mourtzakis M, Zenith L, Myers RP, Abraldes JG, Shaheen AA, Qamar H, Mansoor N, Carbonneau M, Ismond K, Mann S, Alaboudy A, Ma M. A Model to Identify Sarcopenia in Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2016 Oct;14(10):1473-1480.e3. doi: 10.1016/j.cgh.2016.04.040. Epub 2016 May 14. PMID 27189915